CLINICAL TRIAL: NCT06547645
Title: Skilled Nursing Facility at Home Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Baystate Health (Other); UMass Memorial Health (Other); Massachusetts Executive Office of Health and Human Services (EOHHS) (Unknown)
Responsible Party: Principal Investigator, Apurv Soni, Assistant Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00001862
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Skilled Nursing Facility; Rehabilitation; Home Based Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facility-based (No Intervention): Facility based post acute care at a skilled nursing facility, as is the standard care model.
- Home-based (Active Comparator): Home-based Post-Acute Care
  Interventions: Other: Sub-Acute Rehab at Home

INTERVENTIONS:
Other: Sub-Acute Rehab at Home — Patients randomized to the intervention group will receive skilled nursing and rehabilitative care at home upon discharge from the hospital, or when eligible for skilled-nursing facility care when requiring a step up in services at home. Home care will be delivered and overseen by a multidisciplinary clinical team, which will develop individualized care plans based on diagnosis, specific rehabilitation objectives, and broader goals of care.
  Other Names: SNF at Home
  Arms: Home-based

SUMMARY:
Skilled Nursing Facility at Home is a multicenter randomized control trial that aims to evaluate a home-based model of providing post-acute care (PAC). We will enroll 650 hospitalized patients who require rehabilitation and/or skilled-nursing support upon discharge and randomly assign them to an intervention (home-based PAC) or control arm (facility-based PAC). Our design includes two different health systems in Massachusetts: Baystate Health and UMass Memorial Health. We will perform 1:1 randomization between the intervention and control arm using a permuted block design, with stratification by clinical site and payor group. The primary outcome of the trial will be the difference in hospital readmission and mortality rates from the time of enrollment to 30 days after enrollment. Secondary clinical, functional, and cost outcomes include length of stay in PAC, difference in health-related quality of life (HRQoL), and healthcare cost and utilization.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Admitted to an inpatient unit OR receiving home health and requiring an escalation to skilled-nursing facility care
* Require post-acute care in a skilled nursing facility based on the clinical inpatient team's assessment (or, if the participant is coming from home, based on the home health team's assessment)
* Pass the home readiness assessment
* Reside within Greater Worcester or Greater Springfield

Exclusion Criteria:

* Inability to return to a home residence where care can be provided
* Inability for patient or their proxy to provide informed consent for the study
* Requires long-term care
* Requires palliative or hospice care
* On active chemotherapy
* Post-transplant surgery
* Requires hemodialysis
* Requires radiation therapy
* Requires two-person assist or mechanical lift
* Expresses unwillingness to be randomized to SNF OR SNF at Home care
* Considered clinically inappropriate by SNF at Home clinical team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-01-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
30-Day Readmission and Mortality | From time of enrollment to 30 days after enrollment
  Hospital readmission rates and mortality rates between the intervention and control groups in the first 30 days after enrollment

SECONDARY OUTCOMES:
90- and 180- day Readmission and Mortality | From time of enrollment, up to 6 months post-enrollment
  Hospital readmission rates and mortality rates between the intervention and control groups in the 90- and 180- days after enrollment
Days Alive | From time of enrollment, up to 6 months post-enrollment
  Starting with the day of randomization, the total number of days alive outside of the hospital during the study period.
Activities of Daily Living | From time of enrollment, up to 6 months post-enrollment
  Compare the improvement in ability to perform activities of daily living between the intervention and control groups from time of enrollment to 30, 90 and 180-days after enrollment.
Healthcare Costs | From time of enrollment, up to 6 months post-enrollment
  Compare healthcare cost incurred and healthcare utilization between the intervention and control group during the PAC episode as well as from time of enrollment to the end of the PAC episode.
Mortality rate | From time of enrollment to 6 months post-enrollment
  Compare mortality rates during the study period between the intervention and control groups.
Length of stay | From time of enrollment, up to 6 months post-enrollment
  Compare length-of-stay (number of days) that study participants receive post-acute, SNF-level care during the index PAC episode between the intervention and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — University of Massachusetts, Worcester
Locations (2):
- United States (2):
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No